CLINICAL TRIAL: NCT07240077
Title: Beta-lactam Monotherapy Versus Beta-lactam Plus Levofloxacin for the Treatment of Streptococcal Bacteremia: A Multicenter, Randomized, Double-Blind, Pragmatic Trial
Brief Title: Beta-lactam Plus Levofloxacin to Enhance Therapy in Streptococcal Septicemia
Acronym: BLESS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Pinyo Rattanaumpawan, Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 886/2568(IRB3)
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Bacteremia; Streptococcus Infection
Keywords: bacteremia; streptococcus; levofloxacin
MeSH Terms: conditions — Bacteremia; Streptococcal Infections | interventions — beta-Lactams

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beta-lactam monotherapy (Placebo Comparator): Normal saline 150 cc IV drip in 90 minutes once daily for 3-7 days (in a blinding package)
  Interventions: Drug: Beta-lactam monotherapy
- Levofloxacin combination therapy (Experimental): Levofloxacin 750 mg IV drip in 90 minutes once daily for 3-7 days (in a blinding package)
  Interventions: Drug: Beta-lactam plus levofloxacin combination therapy

INTERVENTIONS:
Drug: Beta-lactam monotherapy — Normal saline placebo
  Arms: Beta-lactam monotherapy
Drug: Beta-lactam plus levofloxacin combination therapy — IV Levofloxacin
  Arms: Levofloxacin combination therapy

SUMMARY:
A double-blind randomized controlled trial comparing beta-lactam plus levofloxacin versus beta-lactam monotherapy for the treatment of Streptococcal bacteremia

DETAILED DESCRIPTION:
This randomized, double-blind clinical trial enrolls hospitalized or outpatient adults (≥18 years) with blood cultures positive for Streptococcus spp. who are receiving intravenous beta-lactam monotherapy. Eligible participants continue beta-lactam therapy and are randomized (block size of 4, stratified by site) to receive either intravenous levofloxacin 750 mg once daily or a normal saline placebo for 3-7 days, with dosing adjusted for renal function. The primary outcome is a composite endpoint of unfavorable events, and the secondary outcome is the duration of bacteremia

ELIGIBILITY:
Inclusion Criteria:

1. Adults age>18 years
2. Blood culture positive for Streptococcus (<72 hours before enrollment)

   * at least 1 bottle of S. pyogenes, S. agalactiae, S. pneumoniae, S. suis
   * at least 2 bottle of other Streptococci
3. Receiving or having plan of receiving beta-lactam therapy

Exclusion Criteria:

1. Known allergy to beta-lactam or fluroquinolone antibiotics
2. Pregnancy or lactating mother
3. EKG with QT prolongation
4. Diagnosis of infective endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpointof unfavorable outcome | 28 days after the onset of infection
  a composite endpoint comprising persistent bacteremia lasting more than 5 days, 28-day all-cause mortality, and the development of new metastatic foci within 28 days from infection onset

SECONDARY OUTCOMES:
Duration of bacteremia | 28 days after the onset of infection
  Duration of bacteremia

CONTACTS AND LOCATIONS:
Locations (4):
- Thailand (4):
  - Faculty of Medicine Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Maharaj Nakhon Ratchasima, Nakhon Ratchasima
  - Ratchburi Hospital, Ratchaburi

IPD SHARING:
Plan to Share IPD: No